CLINICAL TRIAL: NCT02754583
Title: Sanitation, Water, and Instruction in Face-washing for Trachoma I/II
Acronym: SWIFT I/II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: The Carter Center (Other); Amhara Public Health Institute (Unknown); Emory University (Other); National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-14004; U10EY023939 (NIH)
Record Dates: First submitted 2015-10-15; First posted 2016-04-28 (Estimated); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Trachoma
Keywords: trachoma; soil transmitted helminths; sanitation; face washing; antibiotics
MeSH Terms: conditions — Trachoma | interventions — Water; Sanitation; Hygiene; Therapeutic Irrigation; Methods; Health; Azithromycin; Tetracycline

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- WASH arm (WUHA) (Experimental): WUHA I, Behavioral: Water, sanitation, and hygiene (WASH) intervention: Communities will receive the water, sanitation, and hygiene (WASH) intervention including community water point construction, hygiene and sanitation education and promotion, community-based hygiene promotion workers, household wash stations, household WASH education books, household soap distribution, and a hygiene curriculum for primary schools.
  WUHA II, Behavioral and Treatment: WASH intervention communities will continue to receive the water, sanitation, and hygiene (WASH) intervention.
  A single mass azithromycin distribution will be given in all 40 WUHA I communities (both intervention and control) after the final study visit (i.e., month 36). Children 6 months and up will be offered azithromycin 20mg/kg; those under 6 months will be offered tetracycline.
  Interventions: Behavioral: Water, sanitation, and hygiene (WASH) intervention; Drug: Azithromycin; Drug: Tetracycline
- Standard of care WASH arm (WUHA) (Other): WUHA I: Standard of care WASH intervention: Communities will continue to receive the standard of care WASH programming offered by the Ethiopian government.
  WUHA II: Standard of care WASH intervention and treatment: Communities will continue to receive the standard of care WASH programming offered by the Ethiopian government.
  A single mass azithromycin distribution will be given in all 40 WUHA I communities (both intervention and control) after the final study visit (i.e., month 36). Children 6 months and up will be offered azithromycin 20mg/kg; those under 6 months will be offered tetracycline.
  These communities will receive a WASH package at the conclusion of the SWIFT II study, including water point construction, hygiene and sanitation promotion, and educational materials.
  Interventions: Behavioral: Standard of care WASH intervention; Drug: Azithromycin; Drug: Tetracycline
- Targeted antibiotics arm (TAITU) (Experimental): Targeted antibiotic treatment: Communities will receive targeted antibiotic treatments for children testing positive for ocular chlamydia at 3, 6, 9, and 12 months after baseline testing. After testing for ocular chlamydia at 12 months, any children testing positive at this time point will receive antibiotic treatments at 15, 18, 21, and 24 months. Children 6 months and up will be offered azithromycin 20mg/kg; those under 6 months will be offered tetracycline.
  Interventions: Drug: Azithromycin; Drug: Tetracycline
- Delayed mass antibiotics arm (TAITU) (Other): Delayed mass antibiotic treatment: Communities will receive no mass azithromycin treatment during the study period. Communities in this treatment group have previously received at least 8 rounds of mass azithromycin treatment. These clusters will be enrolled in an antibiotics treatment program (azithromycin or tetracycline) after the completion of the study.
  Interventions: Other: Control
- Mass antibiotics arm (TAITU) (Active Comparator): Mass antibiotic treatment: Communities will receive mass azithromycin treatment of all individuals aged 6 months and up (20mg/kg for children; 1 g for adults); those younger than 6 months, pregnant, or allergic to macrolide antibiotics will be offered a 2-week course of tetracycline.
  Interventions: Drug: Azithromycin; Drug: Tetracycline

INTERVENTIONS:
Behavioral: Water, sanitation, and hygiene (WASH) intervention — WASH arm: Communities will receive the water, sanitation, and hygiene (WASH) intervention including water point construction and maintenance, hygiene and sanitation education and promotion, community-based hygiene promotion workers, household wash stations, household WASH education books, household soap distribution, and a hygiene curriculum for primary schools.
  Other Names: WASH Upgrades for Health in Amhara (WUHA)
  Arms: WASH arm (WUHA)
Behavioral: Standard of care WASH intervention — Stand of care WASH arm
  Other Names: WUHA
  Arms: Standard of care WASH arm (WUHA)
Drug: Azithromycin — 20mg/kg
  Arms: Mass antibiotics arm (TAITU); Standard of care WASH arm (WUHA); Targeted antibiotics arm (TAITU); WASH arm (WUHA)
Drug: Tetracycline — Tetracycline will be administered in lieu of azithromycin if individual is under 6 months, has a known azithromycin allergy, or is severely ill.
  Arms: Mass antibiotics arm (TAITU); Standard of care WASH arm (WUHA); Targeted antibiotics arm (TAITU); WASH arm (WUHA)
Other: Control — The control group will receive no intervention during the trial. They will be enrolled in mass antibiotic treatment at the conclusion of the trial.
  Arms: Delayed mass antibiotics arm (TAITU)

SUMMARY:
SWIFT I is a series of 3 cluster-randomized trials designed to assess several alternative strategies for trachoma control in communities that have been treated with many years of mass azithromycin distributions. The first trial (named WUHA) compares communities that receive a comprehensive Water, Sanitation, and Hygiene (WASH) package to those that receive no intervention. The second trial (named TAITU-A) compares communities randomized to targeted antibiotic treatment versus those randomized to mass antibiotics for trachoma, and the third trial (TAITU-B) compares communities randomized to targeted antibiotics versus those randomized to delayed antibiotics.

SWIFT II is a continuation of the first trial (WUHA I). WUHA I is an ongoing cluster-randomized trial in rural Ethiopia designed to determine the effectiveness of water, sanitation, and hygiene (WASH) for trachoma. 40 communities were randomized in a 1:1 ratio either to a comprehensive WASH package or to no intervention. The primary outcome is ocular chlamydia, monitored annually for 3 years.

In WUHA II we will treat all 40 WUHA communities with a single mass azithromycin distribution after the month 36 visit, and then continue the WASH intervention only in the 20 communities originally randomized to the WASH arm. We perform annual monitoring visits at months 48, 60, 72, and 84 for the primary outcome of ocular chlamydia among 0-5 year old children. A second aim of WUHA II is to perform a diagnostic test accuracy study of the tests already being conducted as well as several novel tests for trachoma surveillance. The novel tests include inexpensive, point-of-care nucleic acid amplification tests performed on conjunctival swabs, a lateral flow assay for chlamydia seropositivity tested on dried blood spots, and an automated algorithm to detect clinical signs of trachoma from conjunctival photographs. The primary objective of the second aim is to test the sensitivity and specificity of each of these trachoma surveillance tests.

By comparing the combined azithromycin-WASH communities to communities receiving mass azithromycin alone, we investigate the benefit of combining the "A", "F", and "E" components of the SAFE strategy as opposed to focusing on antibiotics alone. This is an important question given the expense of WASH interventions and the limited resources of trachoma programs.

DETAILED DESCRIPTION:
Trachoma is a blinding disease caused by ocular strains of Chlamydia trachomatis. The Carter Center and Proctor Foundation have been jointly conducting trachoma research in the Amhara region of Ethiopia for the past 10 years, through a series of clinical trials. We have found that repeated mass administration of oral azithromycin can greatly reduce the prevalence of trachoma, but mass antibiotics have been unable thus far to eliminate infection.

The World Health Organization recommends not only antibiotics for control of trachoma, but an entire SAFE strategy (Surgery for in-turned eyelids, Antibiotics, Facial hygiene promotion, and Environmental improvements such as latrines and water points). The rationale for the SAFE strategy is based on many years of observational studies on trachoma. Cross-sectional studies have found that clinically active trachoma and ocular chlamydial infection are associated with several indicators of poor hygiene, including dirty faces, face-seeking flies, long distance to water supply, and lack of household latrine. There are few randomized trials testing the impact of WASH improvements on trachoma.

In the past, the WHO has recommended targeted antibiotic treatments to those individuals with active disease, so this could be an alternative treatment strategy that would limit antibiotic use in the community and perhaps be cost-saving. However, little research has assessed targeted treatments as a strategy for trachoma elimination following repeated mass azithromycin distributions.

Our long term goal is to eliminate trachoma even in the most hyperendemic communities. This cluster-randomized clinical trial will determine the role of a comprehensive package of sanitation measures for the elimination of trachoma. We will monitor clinical disease with photography, and monitor infection with a newer chlamydial polymerase chain reaction (PCR) test (Abbott m2000) that is more sensitive than earlier generation tests, and provides quantification. We will monitor other potential health benefits of a WASH intervention and test its overall cost effectiveness. We will also assess a competing strategy for minimizing antibiotic use: that of targeted azithromycin treatments to children testing positive for ocular chlamydia. We will model the long-term cost-effectiveness of these competing strategies for trachoma control after completion of several rounds of mass azithromycin distributions.

Our monitoring has revealed a high uptake of the SWIFT I/WUHA I intervention as well as evidence of subsequent hygiene behavior changes. However, communities started out with a high burden of ocular chlamydia and preliminary data suggests that elimination will be unlikely. We therefore were granted an continuation grant (SWIFT II) to determine the long-term benefit of WASH for trachoma when combined with antibiotics, and second, to explore possibilities for low-cost, highly accurate point-of-care test for chlamydia.

With SWIFT II, we are extending the WUHA I trial by performing a single mass azithromycin distribution in all 40 communities after the final study visit (i.e., month 36), and continuing the WASH intervention in the 20 communities originally randomized to WASH. We are monitoring for ocular chlamydia via PCR of conjunctival swabs. We ask whether antibiotic distributions combined with a comprehensive, well-functioning WASH package is more likely to eliminate trachoma than antibiotics alone. We will also collect extra swabs and dried blood spots during routine monitoring visits and compare several inexpensive, commercially available NAATs and serologic tests for chlamydia. The SWIFT II trial leverages our existing SWIFT I research infrastructure and takes advantage of the fact that the intervention has already been implemented, and will have been operating for more than six years by the end of the proposed study. WASH interventions are thought to take a long time to work given their reliance on changing behavior, and thus we will increase the chances of finding an effect if one truly exists. Moreover, we will advance knowledge regarding trachoma surveillance, which has become increasingly important as the world moves towards global elimination. The results of the SWIFT II study will be of interest to the trachoma community, and regardless of the outcome will directly help trachoma programs decide how to spend their limited resources.

ELIGIBILITY:
Community Level

* Inclusion Criteria

  * Community in a school district that is within the study area of WagHimra
  * Area within each school district with a site identified for water point construction
  * At least 5 rounds of mass azithromycin distributions had been performed within community
* Exclusion Criteria:

  * School districts that are too difficult to reach (more than a 1-day of travel to access)
  * School districts in the 2 urban regions of the study area, since urban communities have better access to water and sanitation and have less trachoma
  * Refusal of village chief

Individual Level

* Inclusion Criteria:

  * All residents residing within a 1.5km radius from the most promising potential water point the water point sites within the school district that were identified for the study
* Exclusion criteria

  * Refusal of participant [or parent/guardian]

Ages: 1 Day to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 47605 (Actual)
Dates: Start 2015-12-05 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Village-specific ocular chlamydia among 0-5 children over time (first trial: WUHA) | 12, 24, 36, 48, 60, 84, 96 months
  Multiple time points will be used in a mixed effects regression model of the village-specific ocular chlamydia prevalences over time in 0-5 year olds as assessed by PCR.
Ocular chlamydia among 8-12 year olds (second trial: TAITU-A) | 24 months
  Cluster-specific prevalence of ocular chlamydia among individuals aged 8-12 years, compared between the targeted azithromycin arm and the mass azithromycin arm.
Incident ocular chlamydia in 0-5 year-olds (third trial: TAITU-B) | 24 months
  Incidence of new ocular chlamydia infection in 0-5 year-olds, compared between the targeted azithromycin arm and the delayed mass azithromycin arm.
Trial-based cost-effectiveness of intervention (intervention costs per percent of chlamydia reduction) | 24 months for TAITU, 36 months for WUHA
  The short term analysis is designed to provide insight into whether each intervention (WASH or targeted antibiotics) is effective for our primary trial outcome of reducing ocular chlamydial infection in children. The time horizon of these analyses will be the duration of each trial.

SECONDARY OUTCOMES:
Quantitative PCR chlamydia load | 12, 24, 36, 48, 60, 84, 96 months
  The analysis is proposed to be identical to that of the ocular chlamydia outcome, except that a village-specific index of chlamydia load at baseline and at follow-up times is used instead of prevalence. The analysis is two-sided at an alpha of 0.05.
  This is a prespecified secondary analysis and will be reported as such.
Follicular trachoma scores; age-stratified (0-5, 6-9, 10 and up for WUHA; 0-5, 8-12 for TAITU) | 12, 24, 36, 48, 60, 84, 96 months
  Follicular trachoma scores (using the 5 level system) will be modeled longitudinally using linear mixed effects regression. Scores are indexed by participant, grader, visit, and village. Participant and village will be modeled as random effects; grader will be modeled as a fixed effect. We will use an AR(1) correlation structure.
Inflammatory trachoma scores; age-stratified (0-5, 6-9, 10 and up for WUHA; 0-5, 8-12 for TAITU) | 12, 24, 36, 48, 60, 84, 96 months
  Inflammatory trachoma grades will be modeled in the same way as Follicular Trachoma.
Clinical trachoma improvement as measured in photography | 12, 24, 36, 48, 60, 84, 96 months
  We anticipate having the following information available. For each child in the sampling frame, we will have a binary improvement score, based on baseline and follow-up photography. We propose to conduct clustered logistic regression (taking into account the clustered nature of the design) using village assignment as the predictor. We will estimate the log odds of the treatment effect. Significance testing will be conducted at 0.05 based on Monte Carlo permutation testing.
Chlamydial load, individual level analysis | 12, 24, 36, 48, 60, 84, 96 months
  Quantitative PCR results at the individual level will be modeled using standard procedures for semi-continuous variables.
Ocular chlamydia; age-stratified (6-9, 10 and up for WUHA; 8-12 for TAITU) | 12, 24, 36, 48, 60, 84, 96 months
  Longitudinal analysis of ocular chlamydia in the age 6-9 group will be modeled at the village level. A similar analysis will consider the 10 and over segment of the population.
Nasopharyngeal pneumococcal macrolide resistance | 12, 24, 36, 96 months
  Using standard microbiological techniques, the lab will process the swabs using media selective for Streptococcus pneumoniae, and then test for antibiotic resistance. Nasopharyngeal macrolide resistance in age 0-5 will be modeled at the village level, using treatment arm as a covariate.
Proportion of the population with clean faces at the village level | 12, 24, 36, 48, 60, 84, 96 months
  The proportion of the population with clean faces will be compared (at the village level) between the two groups, using ANCOVA with baseline values and treatment arm as covariates.
Childhood growth (height) | 12, 24, 36 months
  Longitudinal analysis of anthropometric measurements between the two arms will be conducted using growth curve models.
Childhood growth (weight) | 12, 24, 36 months
  Longitudinal analysis of anthropometric measurements between the two arms will be conducted using growth curve models.
Soil-transmitted helminth prevalence | 12, 24, 36 months
  The prevalence of soil transmitted helminths will be compared between the WUHA treatment arms in a linear mixed effects regression as described above for ocular chlamydia.
Soil-transmitted helminth density | 12, 24, 36 months
  Quantitative soil transmitted helminth results at the individual level will be modeled using standard procedures for semi-continuous variables.
Prevalence of chlamydia and other antigen positivity from serological tests | 12, 24, 36, 48, 60, 84, 96 months
  The prevalence of chlamydia antigen positivity will be compared between the treatment arms in a linear mixed effects regression as described above for ocular chlamydia.
Prevalence of stool-based antigen (diarrheal pathogens, soil transmitted helminths) positivity from serological tests | 12, 24, 36, 48, 60, 84, 96 months
  The prevalence of soil transmitted helminths will be compared between the treatment arms in a linear mixed effects regression as described above for ocular chlamydia.
Intestinal microbiome from rectal sample | 24 months
  Intestinal microbiome from rectal sample, using 16S rRNA deep sequencing and/or next generation sequencing
Sensitivity and specificity of detecting STH using rectal swabs | 24 months
  Sensitivity and specificity of detecting STH using rectal swabs with logistic mixed-effects. Bulk stool samples will be used as the gold standard.

CONTACTS AND LOCATIONS:
Overall Officials: Zerihun Tadese, MD, MPH, Study Director — The Carter Center Ethiopia; Jeremy D Keenan, MD, MPH, Principal Investigator — University of California San Francisco Proctor Foundation; Dionna M Wittberg, MPH, Study Director — UCSF Proctor Foundation
Locations (1):
- The Carter Center Ethiopia, Addis Ababa, Ethiopia

REFERENCES:
- [Derived] Wittberg DM, Admassu F, Aragie S, Dagnew A, Hailu D, Tadesse Z, Zeru T, Thompson IJB, Abdu S, Beyecha S, Birhanu T, Getachew H, Getnet B, Kabtu E, Shibiru M, Tekew S, Wondimteka B, Freeman MC, Nash SD, Lietman TM, Keenan JD. The Effect of a Water, Sanitation, and Hygiene Intervention on Clinical Trachoma: A Cluster-Randomised Trial. Trop Med Int Health. 2026 Jan 18. doi: 10.1111/tmi.70086. Online ahead of print. PMID 41548574
- [Derived] Frank T, Thompson IJB, Aragie S, Wittberg DM, Tadesse W, Dagnew A, Hailu D, Melo JS, Zeru T, Tadesse Z, Arnold BF, Freeman MC, Nash SD, Callahan EK, Porco TC, Lietman TM, Keenan JD. Effect of water, sanitation, and hygiene on childhood growth in Ethiopia: a cluster-randomized trial. Int J Hyg Environ Health. 2026 Jan;271:114718. doi: 10.1016/j.ijheh.2025.114718. Epub 2025 Nov 27. PMID 41314021
- [Derived] Caleon RL, Admassu F, Aragie S, Hailu D, Dagnew A, Zeru T, Wittberg DM, Thompson IJB, Abdu S, Beyecha S, Birhanu T, Getachew H, Getnet B, Kabtu E, Shibiru M, Tekew S, Wondimteka B, Lietman TM, Nash SD, Freeman MC, Keenan JD. Photographic grading to evaluate facial cleanliness and trachoma among children in Amhara region, Ethiopia. PLoS Negl Trop Dis. 2024 Jul 11;18(7):e0012257. doi: 10.1371/journal.pntd.0012257. eCollection 2024 Jul. PMID 38991011
- [Derived] Tedijanto C, Aragie S, Gwyn S, Wittberg DM, Zeru T, Tadesse Z, Chernet A, Thompson IJB, Nash SD, Lietman TM, Martin DL, Keenan JD, Arnold BF. Seroreversion to Chlamydia trachomatis Pgp3 Antigen Among Children in a Hyperendemic Region of Amhara, Ethiopia. J Infect Dis. 2024 Aug 16;230(2):293-297. doi: 10.1093/infdis/jiad602. PMID 38134305
- [Derived] Aragie S, Wittberg DM, Tadesse W, Dagnew A, Hailu D, Chernet A, Melo JS, Aiemjoy K, Haile M, Zeru T, Tadesse Z, Gwyn S, Martin DL, Arnold BF, Freeman MC, Nash SD, Callahan EK, Porco TC, Lietman TM, Keenan JD. Water, sanitation, and hygiene for control of trachoma in Ethiopia (WUHA): a two-arm, parallel-group, cluster-randomised trial. Lancet Glob Health. 2022 Jan;10(1):e87-e95. doi: 10.1016/S2214-109X(21)00409-5. PMID 34919861
- [Derived] Wittberg DM, Aragie S, Tadesse W, Melo JS, Aiemjoy K, Chanyalew M, Emerson PM, Freeman MC, Nash SD, Callahan EK, Tadesse Z, Zerihun M, Porco TC, Lietman TM, Keenan JD. WASH Upgrades for Health in Amhara (WUHA): study protocol for a cluster-randomised trial in Ethiopia. BMJ Open. 2021 Feb 22;11(2):e039529. doi: 10.1136/bmjopen-2020-039529. PMID 33619183

DOCUMENTS (2):
  • Study Protocol (2022-03-04): https://cdn.clinicaltrials.gov/large-docs/83/NCT02754583/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-19): https://cdn.clinicaltrials.gov/large-docs/83/NCT02754583/SAP_001.pdf